CLINICAL TRIAL: NCT03491371
Title: The Effectivity and Toxicity of Methylsulfonic Apatinib for Extensively Pre-treated Advanced Sarcoma: a Multicentric Retrospective Study in China
Brief Title: Apatinib for Advanced Sarcoma: Results From Multiple Institutions' Off-label Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 01
Record Dates: First submitted 2018-03-31; First posted 2018-04-09 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Efficacy; Toxicity
Keywords: apatinib; tyrosine-kinase inhibitors; osteosarcoma; Ewing sarcoma; chondrosarcoma; soft-tissue sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Chondrosarcoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- osteosarcoma (Experimental): all patients had been given apatinib alone
  Interventions: Drug: Methylsulfonic apatinib
- Ewing sarcoma (Experimental): Some of patients had been given apatinib alone while some of them had been given apatinib+everolimus
  Interventions: Drug: Methylsulfonic apatinib
- soft tissue sarcoma (Experimental): Some of the patients had been given apatinib alone while some of the patients had been given apatinib together with GT chemotherapy, which was gemcitabine 1000 mg/m2 d1,8 and docetaxel 75 mg/m2 d8 once every 21 day.
  Interventions: Drug: Methylsulfonic apatinib
- Chondrosarcoma (Experimental): Patients were given apatinib alone
  Interventions: Drug: Methylsulfonic apatinib

INTERVENTIONS:
Drug: Methylsulfonic apatinib — Anti-angiogenesis Tyrosine kinase inhibitor which specifically inhibits VEGFR-2.

SUMMARY:
Anti-angiogenesis Tyrosine kinase inhibitors (TKIs) have been proved to show promising effects on prolonging progression-free survival (PFS) for advanced sarcoma after failure of standard multimodal Therapy. Methylsulfonic apatinib is one of those TKIs which specifically inhibits VEGFR-2. This study summarizes the experience of three Peking University affiliated hospitals in off-label use of apatinib in the treatment of extensively pre-treated sarcoma.

DETAILED DESCRIPTION:
The investigators retrospectively analysed files of patients with advanced sarcoma not amenable to curative treatment, who were receiving an apatinib-containing regimen between June 1, 2015 and December 1, 2016. Fifty-six patients were included: 22 osteosarcoma, 10 Ewing's sarcoma, 3 chondrosarcoma and 21 soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed high-grade sarcoma;
* 2) initial treatment in the orthopedic oncology departments of the three affiliated hospitals of Peking University;
* 3) tumors not amenable to curative treatment or inclusion in clinical trials;
* 4) unresectable local advanced lesions or multiple metastatic lesions that could not be cured by local therapy;
* 5) measurable lesions according to Response Evaluation Criteria for Solid Tumors (RECIST1.1) [8];
* 6) Eastern Cooperative Oncology Group performance status 0 or 1 [9]; and 7) acceptable hematologic, hepatic, and renal function.

Exclusion Criteria:

* had been previously exposed to other TKIs;
* had central nervous system metastasis;
* had other kinds of malignant tumors at the same time; had cardiac insufficiency or arrhythmia;
* had uncontrolled complications such as diabetes mellitus, coagulation disorders, urine protein ≥ ++ and so on;
* had pleural or peritoneal effusion that needs to be handled by surgical treatment;
* combined with other infections or wounds
* were pregnant or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
objective response rate | 3 month
  CR+PR accroding to RECIST 1.1

SECONDARY OUTCOMES:
progression-free survival, PFS | 4 months and 6 months
  PFS was defined as time from the start of using apatinib until disease progression or death, whichever occurred first.
duration of response, DOR | 4 months
  The time from appearance of response or stable disease to progression or death was thus considered the DOR
Overall Survival,OS | 12 months
  OS was defined as time from the start of using apatinib until death.
toxicity | 12 months
  accroding to the Common Terminology Criteria for Adverse Events 4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Musculoskeletal Tumor Center of Peking University People's Hospital, Beijing
  - Peking University Shougang Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No